CLINICAL TRIAL: NCT02682342
Title: Hyperglycemia and Mitochondrial Function in The Endothelium of Humans
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Michael E. Widlansky, Associate Professor of Medicine, Medical College of Wisconsin
Other Study IDs: PRO26013
Record Dates: First submitted 2016-02-08; First posted 2016-02-15 (Estimated); Results first posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-11

CONDITIONS: Diabetes; Hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus; Hyperglycemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples and endothelial cells obtained will be saved for banking for future studies as possible.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy Subjects: Healthy subjects meeting inclusion criteria will be administered a 75 g glucose solution one time (orally). Subjects will be ages 21-70 years with no evidence of diabetes, hypertension, metabolic syndrome, or high cholesterol at the time of screening. Potential subjects with a history of atherosclerotic disease, chronic renal insufficiency (plasma creatinine > 1.5 men, > 1.5 women), liver enzymes > 2.5x normal, pregnant at the time of screening will be excluded
  Interventions: Other: 75 g glucose solution

INTERVENTIONS:
Other: 75 g glucose solution — This is the same as the standard oral glucose challenge dose and route given clinically

SUMMARY:
In this study, the investigators will test the hypothesis that acute in vivo exposure to hyperglycemia increases mitochondrial network fragmentation and mitochondrial reactive oxygen species production (ROS) production in human arterial endothelial cells.

DETAILED DESCRIPTION:
Subjects will be recruited according to our inclusion/exclusion criteria. The investigators employ a multifaceted approach to recruitment, including flyers, community newspaper ads, internet ad postings, and direct recruitment from the Internal Medicine Clinics of Froedtert Memorial Lutheran Hospital/Medical College of Wisconsin which saw approximately 50,000 unique outpatient visits over last year. The electronic health record is leveraged to identify potential subjects by HIPAA guidelines and Medical College of Wisconsin policies. Potential subjects will undergo phenotyping that includes a detailed medical history, anthropomorphic measurements, blood pressure and heart rate measurements, and a blood draw for measurements that include fasting lipids, glucose, and glycosylated hemoglobin, creatinine, and liver function tests. Healthy, non-DM subjects who pass the screening as per the inclusion/exclusion criteria in Table 2 will be enrolled in the study protocol.

Following an overnight fast (12 hours), subjects will come in the morning to our Adult Translational Research Unit (A-TRU) which is part of the Clinical Translational Research Initiative of Southeast Wisconsin (8UL1TR000055). An antecubital intravenous line will be placed to facilitate blood glucose sampling during the hyperglycemic challenge. An antecubital intravenous catheter will be placed to facilitate obtaining endothelial cells from the vein by J-wire biopsy for of mitochondrial testing. The principal investigator has published experience with the J-wire endothelial cell biopsy technique, and the technique has been extensively validated technique. An initial venous glucose sample will be taken from the antecubital vein and an initial J-wire biopsy of the radial artery endothelium will be performed through the radial arterial line. Subjects will then be asked to drink a standardized 75 g glucose drink created by the A-TRU nutritionist- a standard oral glucose challenge as used clinically. Blood glucose samples will be taken hourly after that until 4 hours post drink ingestion. At one and 4 hours post-ingestion, J-wire endothelial biopsies of the radial artery will be repeated. Four separate J wires will be passed into the radial artery for each measurement time point (0,1, and 4 hours).

In non-diabetic subjects, the 75 g oral challenge induces a peak increase in systemic glucose at 1-hour post-administration at which time endothelial dysfunction is concomitantly detectable. Endothelial cells will be obtained via J-wire capture technique. A portion of the endothelial cells isolated from the J-wires will be used to measure mitochondrial network complexity prior hyperglycemic challenge, 1-hour post challenge, and 4 hours post challenge. The investigators will visualize the mitochondrial networks in these cells using our previously reported and validated immunofluorescence method using cytochrome c antibodies to tag the mitochondria. Network fragmentation (high number=greater fragmentation and fission) will be quantified by network fragmentation count calculated with ImageJ (NIH, Bethesda) using a validated protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Adult age 21 to 70
2. No evidence of metabolic syndrome or diabetes, hypertension (BP≥140/90), or high cholesterol (LDL≥160) at the time of screening.

Exclusion Criteria:

1. History of stroke, peripheral arterial disease, or coronary artery disease (as defined by the presence of at least one coronary stenosis ≥ 40% on angiography or by confirmed history of myocardial infarction by standard criteria).
2. History of bleeding disorders.
3. Evidence of other evident major illness including chronic renal insufficiency (plasma creatinine > 1.4 for women or 1.5 for men), liver disease (liver enzymes greater than 2.5 x normal), and cancer
4. currently undergoing therapy or had therapy for cancer within 1 year of enrollment.
5. Pregnancy as determined by urinary human chorionic gonadotropin beta test
6. Thienopyridine, anti-thrombin/Xa, or warfarin therapy at time of screening
7. On medication for cholesterol or blood pressure

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects without evidence of diabetes, insulin resistance, hypertension, or elevated cholesterol. Subjects will also be without prevalent cardiovascular disease, chronic renal insufficiency, or chronic liver disease.
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2016-03-09 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Micahel E Widlansky, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
The data may be available to qualified investigators following study completion and initial publication of the data with collaboration with the study PI.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment in southeastern Wisconsin by flyers and electronic advertisements from November 2016 through December 2019
Pre-assignment Details: Four subjects were disqualified during screening for cardiovascular risk factors (3 due to elevated total cholesterol and one due to hypertension). One additional subject withdrew consent during screening. One additional subject qualified for the study but never scheduled a study visit. These subjects are not in the 35 subject considered enrolled in the study
Period: Overall Study
Arm/Group | Healthy Subjects
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Subjects
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 27
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 35
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 26.6 (4.3)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 118 (10)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 72 (7)
Hemoglobin A1C [Mean (Standard Deviation); unit: %] | 5.4 (0.4)
Heart Rate [Mean (Standard Deviation); unit: bpm] | 70 (11)
Total Cholesterol [Mean (Standard Deviation); unit: mg/dl] | 183 (35)
HDL Cholesterol [Mean (Standard Deviation); unit: mg/dl] | 63 (21)
LDL Cholesterol [Mean (Standard Deviation); unit: mg/dl] | 106 (26)
Triglycerides [Mean (Standard Deviation); unit: mg/dl] | 71 (28)
Fasting Glucose [Mean (Standard Deviation); unit: mg/dl] | 93 (9)
Serum Creatinine [Mean (Standard Deviation); unit: mg/dl] | 0.88 (0.18)
Waist Circumference [Mean (Standard Deviation); unit: cm] | 91 (13)

OUTCOME MEASURES:

1. Primary Outcome: Change in Mitochondrial Network Complexity of Endothelial Cells as Measured by Mitochondrial Network Fragment Ratio
Description: The investigators visualize the mitochondrial network complexity in these cells using our previously reported and validated immunofluorescence method using cytochrome c antibodies to tag the mitochondria. Network fragmentation (total number of fragments/ total fluorescent pixels*100) will be quantified by network fragmentation count calculated with ImageJ (NIH, Bethesda) using a validated protocol.
Time Frame: Measured at 0,1, and 2 hours after administration
Population: The samples quality when we went back to look at the cells was too poor to obtain valid and reproducible measurements so the outcome was not used.
Arm/Group | Healthy Subjects
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the patient enrollment period of the study (from 2016 through 2023). Each subject was only followed for adverse events for 2 hours following the completion of study protocol
Description: Asymptomatic hypoglycemia
Arm/Group | Healthy Subjects
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 4/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Healthy Subjects (N=35)
Asymptomatic hypoglycemia (Metabolism and nutrition disorders) | 4 — Asymptomatic blood sugars were detected at 2 hours (blood glucose < 60 mg/day) in 4 patients on protocol. These were treated with allowing the patient to drink juice and eat.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-09-04): https://cdn.clinicaltrials.gov/large-docs/42/NCT02682342/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-20): https://cdn.clinicaltrials.gov/large-docs/42/NCT02682342/ICF_001.pdf